CLINICAL TRIAL: NCT04379037
Title: Vagus Nerve Stimulation ARDS Prevention Trial for COVID-19 Hospitalized Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemechek Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCM-001
Record Dates: First submitted 2020-05-05; First posted 2020-05-07 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Severe Acute Respiratory Syndrome Coronavirus 2
Keywords: vagus nerve stimulation; COVID-19; Acute Respiratory Distress Syndrome
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: The objective of this study is to determine the therapeutic effect of transcutaneous vagus nerve stimulation in patients with moderate, severe or critical pneumonia associated with Coronavirus Disease 2019 (COVID-19).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Arm (Experimental): Adults over 18 years of age hospitalized because of COVID-19 infection will be treated with transcutaneous auricular vagus nerve stimulation (taVNS).
  Interventions: Device: Transcutaneous Auricular Vagus Nerve Stimulation

INTERVENTIONS:
Device: Transcutaneous Auricular Vagus Nerve Stimulation — Transcutaneous vagus nerve stimulation involves stimulating the auricular branch of the vagus nerve with a imperceptible electrical current within the concha of the ear.

SUMMARY:
This trial is designed to determine if the inflammation modulating effect of vagus nerve stimulation can improve pulmonary function and limit progression to ARDS in hospitalized COVID-19 hospitalized patients.

DETAILED DESCRIPTION:
Patients hospitalized with COVID-19 predominantly die of organ failure due to a surge of pro-inflammatory cytokines triggering the need for mechanical ventilation, often due to acute respiratory distress syndrome (ARDS). Known as a cytokine storm, the surge in cytokines is similar to the excessive inflammatory reaction associated with septic shock.

Anti-viral agents will most likely be required to reduce the molecular viral burden in COVID-19 patients, but an additional approach to control the damaging cytokine release is required to alter the course of disease in hospitalized patients and improve chances of survival. Immunosuppressant drugs may reduce inflammation and the tissue damaging cytokines, but they could also be detrimental by inhibiting natural anti-viral immune responses (i.e., suppression of interferons), thereby delaying viral clearance and increasing the risk of secondary infections and death.

The reason for the severity of the disease course in some individuals may lie in the regulation of the immune system by the vagus nerve. The vagus nerve is involved in an inflammation controlling reflex similar to the blood pressure regulating baroreflex. The vagus inflammatory reflex is triggered when the afferent vagus nerve senses inflammatory products through peripheral receptors.

Vagus nerve activity is relayed through the central nervous system to the efferent vagus nerve. This pathway involves the splenic nerve, which when activated releases norepinephrine and results in suppression of pro-inflammatory cytokine production by macrophages and alleviates inflammation in many pathological settings (e.g., endotoxemia, peritonitis, or acute kidney injury).

Electrical stimulation of the vagus nerve using VNS can improve the body's natural ability to regulate the inflammatory response and may be potent enough to suppress pro-inflammatory cytokines and prevent death from COVID-19, especially if used early enough in the course of hospitalization.

In rat models of sepsis, VNS attenuates the release of pro-inflammatory cytokines, prevents hypotension, modulates coagulation, and prevents fibrinolysis activation, decreasing organ dysfunction, and improving survival. Human studies also demonstrate that VNS suppresses the production of pro-inflammatory cytokines and improves clinical symptoms in rheumatoid arthritis, intractable epilepsy, atrial fibrillation, and Crohn's Disease.

This suggests that VNS may be effective in treating disorders characterized by cytokine dysregulation and that it has the potential to prevent hospitalized patients with COVID-19 from progressing to respiratory failure and death.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who are 18 years of age
2. Tested positive or suspected/presumed positive for COVID-19 infection
3. Patients requiring hospital admission moderate to severe pneumonia and pneumopathy
4. Patients showing fever and respiratory symptoms with radiological findings of pneumonia
5. Respiratory distress (≧30 breaths/ min) or Oxygen saturation ≤93% at rest in ambient air; or oxygen saturation ≤97 % with O2 > 5L/min
6. Patient is able to provide signed and witnessed Informed Consent

Exclusion Criteria:

1. Already enrolled in a trial for COVID-19 therapy
2. Potentially life threatening heart rhythm
3. Pregnancy or potential pregnancy
4. Current implantation of an electrical and/or neurostimulator device, including but not limited to a cardiac pacemaker or defibrillator, vagal neurostimulator, deep brain stimulator, spinal stimulator, bone growth stimulator, or cochlear implant
5. History of aneurysm, intracranial hemorrhage, brain tumors, or significant head trauma
6. Belongs to a vulnerable population or has any condition such that his or her ability to provide informed consent, comply with the follow-up requirements, or provide self-assessments is compromised (e.g. homeless, developmentally disabled and prisoner)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-06-27 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-11-01 (Actual)

PRIMARY OUTCOMES:
Survival without need of mechanical ventilation | Day 14 since symptom onset
  Survival
Cumulative incidence of successful tracheal extubation at day 14 since symptom onset. | Day 14 since symptom onset
  Successful tracheal extubation

SECONDARY OUTCOMES:
Survival at day 14 of hospitalization | Day 14
  Survival
Duration of hospitalization | Day 28
  Duration of hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Zonal Virgen del Carmen de Zárate, Zárate, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehta P, McAuley DF, Brown M, Sanchez E, Tattersall RS, Manson JJ; HLH Across Speciality Collaboration, UK. COVID-19: consider cytokine storm syndromes and immunosuppression. Lancet. 2020 Mar 28;395(10229):1033-1034. doi: 10.1016/S0140-6736(20)30628-0. Epub 2020 Mar 16. No abstract available. PMID 32192578
- [Background] Kaniusas E, Kampusch S, Tittgemeyer M, Panetsos F, Gines RF, Papa M, Kiss A, Podesser B, Cassara AM, Tanghe E, Samoudi AM, Tarnaud T, Joseph W, Marozas V, Lukosevicius A, Istuk N, Sarolic A, Lechner S, Klonowski W, Varoneckas G, Szeles JC. Current Directions in the Auricular Vagus Nerve Stimulation I - A Physiological Perspective. Front Neurosci. 2019 Aug 9;13:854. doi: 10.3389/fnins.2019.00854. eCollection 2019. PMID 31447643
- [Background] Tanaka S, Hammond B, Rosin DL, Okusa MD. Neuroimmunomodulation of tissue injury and disease: an expanding view of the inflammatory reflex pathway. Bioelectron Med. 2019 Aug 13;5:13. doi: 10.1186/s42234-019-0029-8. eCollection 2019. PMID 32232102
- [Background] Chen G, Wu D, Guo W, Cao Y, Huang D, Wang H, Wang T, Zhang X, Chen H, Yu H, Zhang X, Zhang M, Wu S, Song J, Chen T, Han M, Li S, Luo X, Zhao J, Ning Q. Clinical and immunological features of severe and moderate coronavirus disease 2019. J Clin Invest. 2020 May 1;130(5):2620-2629. doi: 10.1172/JCI137244. PMID 32217835